CLINICAL TRIAL: NCT05645614
Title: Retrospective Evaluation of Pain and Anxiety in Standard Routine Care During Abortion Under Local Anesthesia, in an Abortion Center
Brief Title: Anxiety and Pain During Intervention for Abortion Under Local Anesthesia
Acronym: ADIAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220368
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Abortion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: EVALUATION OF PAIN — PAIN EVALUATION THANKS TO SCALES

SUMMARY:
The aim of the study is to retrospectively analyze pain and anxiety assessment data previously collected in routine care in women who had an abortion under local anesthesia in order to identify the predictive factors of pain and anxiety, as well as to compare the results with previously published data. The participants are women who underwent abortion under local anesthesia in the gynecology department of the Pitié Salpêtrière Hospital between May and October 2021.

DETAILED DESCRIPTION:
Voluntary interruption of pregnancy corresponds to a social demand. The French National Authority for Health recommends that any woman wishing to have a surgical abortion should have the choice between general anesthesia and local anesthesia. The advantages of local anesthesia are its simplicity and safety; the disadvantages are that the state of consciousness during the procedure may be associated with anxiety, and the perception of persistent pain despite the local anesthesia.

The majority of patients express pain during the procedure. Anxiety may be a major predictor of pain during the procedure. Moreover, beyond its possible involvement in pain, anxiety is also a factor of patient discomfort in its own right.

The 10-point verbal numerical scale was used for assessing pain and anxiety. The State Trait Anxiety Inventory (STAI), a 20-item anxiety scale, is also used as a reference to measure anxiety. This scale is carried out for patients undergoing an abortion under local anesthesia in the department.

Other factors could have an impact on the level of pain : age, pregnancy term, parity, history of dysmenorrhea, history of domestic violence or sexual violence.

The investigator team conduct a retrospective analysis in a cohort of patients who underwent an abortion under local anaesthesia in the obstetrics gynecology department of La Pitié Salpêtrière, analyzing their level of pain before, during and after the intervention The secondary objective is to analyze their anxiety level. Age, term of pregnancy, parity, history of dysmenorrhea, history of violence will be analyzed as potential predictive factors of pain.

ELIGIBILITY:
Inclusion Criteria:

* patients who need an abortion under local anesthesia
* Women who speak and read French

Exclusion Criteria:

* NA

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who had an abortion under local anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Pain level of the patient before, during and after (10min post surgery) the abortion procedure under local anesthesia. | 3 hours
  Evolution of pain over time (from preoperative to postoperative), self-assessed on a numerical scale from 0 to 10

SECONDARY OUTCOMES:
Anxiety level of the patient before, during and after (10min post surgery) the abortion procedure under local anesthesia. | 3 hours
  Evolution of Anxiety over time (from preoperative to postoperative), self-assessed on a numerical scale from 0 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié Salpetrière, Paris, France

IPD SHARING:
Plan to Share IPD: No